CLINICAL TRIAL: NCT04606758
Title: Randomized Controlled Trial Comparing Surgical Outcomes Following PCNL Under Ultrasound Control and PCNL Under Fluoroscopic Control in the Treatment of Kidney Stones
Brief Title: Fluoroscopic Guided vs US-guided Percutaneous Nephrolithotripsy for the Treatment of Stone Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Astana Medical University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8
Record Dates: First submitted 2020-10-15; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Urolithiasis; Kidney Stone; Kidney Diseases; Ureteral Calculi; Kidney Calculi
MeSH Terms: conditions — Urolithiasis; Kidney Calculi; Kidney Diseases; Ureteral Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCNL under fluoroscopic control (Active Comparator)
  Interventions: Procedure: PCNL under fluoroscopic control
- PCNL under ultrasound control (Active Comparator)
  Interventions: Procedure: PCNL under ultrasound control

INTERVENTIONS:
Procedure: PCNL under fluoroscopic control — Patients receive standard of care treatment for their urolithiasis using standard PCNL under fluoroscopic guidance
  Arms: PCNL under fluoroscopic control
Procedure: PCNL under ultrasound control — Patients receive standard of care treatment for their urolithiasis using standard PCNL under US guidance
  Arms: PCNL under ultrasound control

SUMMARY:
Randomized comparison of patient outcomes following fluoroscopic guided PCNL versus ultrasound-guided PCNL.

DETAILED DESCRIPTION:
This study is a randomized controlled trial that compares the operative outcomes and complications of fluoroscopic guided-percutaneous nephrolithotomy versus ultrasound-guided PCNL for renal stones. This study will be a prospective randomized controlled clinical trial with patients who have already agreed to undergo PCNL. Patients will be randomized at a 1:1 ratio to receive either PCNL under fluoroscopic guidance or PCNL under ultrasound guidance. Patients will be asked to complete pre-operative, and postoperative quality of life questionnaires, and to allow the collection of one additional vial of blood for measurement of factors associated with inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for PCNL at participating institution
* Patients of all ethnic backgrounds
* Stone size over 10 mm in diameter and a density over 900 Hounsfield units
* Patients with a large calculus in the upper third of the ureter

Exclusion Criteria:

* Pregnancy
* infectious disease of the genitals;
* conditions that violate the configuration of the kidneys (curvature of the spinal column)
* anomalies in the development of the kidneys with impaired configuration and position of the kidneys (horseshoe kidney, bisque kidney, S-shaped kidney, L-shaped kidney, lumbar dystopia, iliac dystopia, pelvic dystopia)
* presence of nephrostomy drainage in the target kidney;
* urethral stricture or other reason leading to the inability to carry out ureteral catheterization;
* other conditions that are contraindications to surgical treatment, such as uncontrolled diabetes mellitus, acute cardiovascular conditions, liver failure, alcoholism, and drug addiction;
* patients who are unable to understand the purpose of the study or refuse further follow-up observation and instructions after treatment;
* patients with a history of mental illness;
* participation in another research that interferes with this research;
* acute renal failure;
* dissecting aortic aneurysm;
* acute hypertensive encephalopathy;
* heavy arterial bleeding;
* myocardial infarction less than six months before enrollment in the study;
* Stroke less than six months before enrollment in the study;
* Insufficiency of blood circulation III-IV New York Heart Association class;
* Severe rhythm and conduction disturbances;
* Increase in the level of liver transaminases by more than three times;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Blood loss as estimated by postoperative decreases in haemoglobin | Post-operative day 1

SECONDARY OUTCOMES:
Surgical outcomes | 6 months
  Outcome measures by using the clavien dindo classification system
Asses the easiness of accessibility of the targeted stone | Intraoperatively
  Outcome measures by counting numbers of puncture trial
The Puncture fluoroscopy screening time | Intraoperatively
  assessed on the monitor of C-Arm.

IPD SHARING:
Plan to Share IPD: Undecided